CLINICAL TRIAL: NCT01726413
Title: A Phase II, 4-Week Randomised, Double-Blind, Parallel Group, Placebo Controlled Proof of Concept Study to Evaluate Efficacy, Safety and Tolerability of GRC 17536 in Patients With Painful Diabetic Peripheral Neuropathy.
Brief Title: A Clinical Trial to Study the Effects GRC 17536 in Patients With Painful Diabetic Peripheral Neuropathy (Painful Extremities Due to Peripheral Nerve Damage in Diabetic Patients).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Collaborators: Glenmark Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRC 17536-203; 2012-002320-33 (EudraCT Number)
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Painful Diabetic Peripheral Neuropathy
Keywords: Diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Arm (Experimental): GRC17356 for daily administration
  Interventions: Drug: GRC 17356
- Placebo (Placebo Comparator): Matching placebo for daily administration
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: GRC 17356
  Arms: Test Arm
Drug: Matching Placebo
  Arms: Placebo

SUMMARY:
Diabetic peripheral neuropathy (DPN) represents a diffuse symmetric and length-dependent injury to peripheral nerves that has major implications on quality of life (QOL), morbidity, and costs from a public health perspective. Painful diabetic neuropathy affects approximately 16% of patients with diabetes. Pharmacological agents used in the management of painful DPN mainly include tricyclic antidepressants, selective serotonin and norepinephrine reuptake inhibitors, opioid, and anti epileptic drugs. The available treatment options do not give total relief, are not effective in all patients, and only about one-third of patients may achieve more than 50% pain relief. Hence newer therapies are required for the treatment of DPN. The primary outcome measures will be the change from baseline to end of treatment in the mean 24-hour average pain intensity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to provide voluntary written informed consent
2. Male and female patients ≥18 yrs and ≤75 yrs
3. Patients with diabetes mellitus with painful peripheral neuropathy for at least 6 months
4. A baseline 24-hour average daily pain intensity score ≥5
5. Women must be of non child-bearing potential, defined as post menopausal or surgically sterile

Exclusion Criteria:

1. Other chronic pain conditions not associated with DPN, that may confound the assessment of neuropathic pain
2. Other causes of neuropathy or lower extremity pain
3. Complex regional pain syndrome or trigeminal neuralgia
4. Lower extremity amputations other than toes
5. Participation in another study with an investigational compound within the previous 90 days prior to study medication administration, or concurrent participation in another clinical study
6. Major depression.
7. Presence or history of cancer within the past 5 years with the exception of adequately treated localized basal cell skin cancer or in situ uterine cervical cancer.
8. Patients with clinically significant or uncontrolled hepatic, gastrointestinal, cardiovascular, respiratory, neurological (other than neuropathy), psychiatric, hematological, renal, or dermatological disease, or any other medical condition that according to Investigator's medical judgment: Could interfere with the accurate assessment of safety or efficacy, or, Could potentially affect a patient's safety or study outcome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Mean 24-hour average pain intensity (API) score. | Week 4

SECONDARY OUTCOMES:
Mean night-time API Score | 4 weeks
Patient Global Impression of Change | 4 weeks
Clinician Global Impression of Change | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Balamurugan Ramanathan, Principal Investigator — Kovai Diabetes Speciality Centre and Hospital; Dr. Vijay Viswanathan, Principal Investigator — MV Hospital for Diabetes (P) Ltd; Dr. Mallikarjun V Jali, Principal Investigator — K.L.E.S Dr. Prabhakar Kore Hospital & Medical research Centre; Dr. Sunil M Jain, Principal Investigator — TOTALL Diabetes Hormone Institute; Dr. Dinesh Dhanwal, Principal Investigator — Maulana Azad Medical College & Associate Hospitals; Dr. S Srikanta, Principal Investigator — Jnana Sanjeevani Medical Centre; Dr. Jayashri Shembalkar, Principal Investigator — Getwell Hospital and Research Centre; Dr Peter Dewland, Principal Investigator — ICON Manchester CPU; Dr. Prof Thomas Forst, Principal Investigator — Institute for Clinical Research and Development( IKFE-CRO GmbH BahnhofstraBe 8A); Dr. Paramesh Shammana, Principal Investigator — Bangalore Clinisearch; Dr. Arthur Asirvatham, Principal Investigator — Arthur Asirvathma Hospital; Dr. Mohan Magdum, Principal Investigator — Jehangir Clinical Development Centre Pvt. Ltd.; Dr. Blanka Lubenova, Principal Investigator — NeuroHelp s.r.o; Dr. David Dolezil, Principal Investigator — DADO Medical s.r.o
Locations (15):
- Czechia (3):
  - NeuroHelp s.r.o, Olomouc, Prague
  - DADO Medical s.r.o, Prague, Prague
  - DADO Medical s.r.o, Říčany, Ricany
- Institute for Clinical Research and Development( IKFE-CRO GmbH BahnhofstraBe 8A), Mainz, Germany, Germany
- India (10):
  - Bangalore Clinisearch, Bangalore, Karnataka
  - K.L.E.S Dr. Prabhakar Kore Hospital & Medical research Centre, Belagavi, Karnataka
  - Jnana Sanjeevani Medical Centre, Bangalore, Karntaka
  - TOTALL Diabetes Hormone Institute, Indore, Madhya Pradesh
  - Getwell Hospital and Research Centre, Nagpur, Maharashtra
  - Jehangir Clinical development Centre Pvt Ltd, Pune, Maharashtra
  - Maulana Azad Medical College & Associate Hospitals, New Delhi, New Delhi
  - MV Hospital for Diabetes (P) Ltd, Chennai, Tamil Nadu
  - Kovai Diabetes Speciality Centre and Hospital, Coimbatore, Tamil Nadu
  - Arthur Asirvathma Hospital, Madurai, Tamil Nadu
- ICON Manchester CPU, Manchester, UK, United Kingdom

REFERENCES:
- [Derived] Jain SM, Balamurugan R, Tandon M, Mozaffarian N, Gudi G, Salhi Y, Holland R, Freeman R, Baron R. Randomized, double-blind, placebo-controlled trial of ISC 17536, an oral inhibitor of transient receptor potential ankyrin 1, in patients with painful diabetic peripheral neuropathy: impact of preserved small nerve fiber function. Pain. 2022 Jun 1;163(6):e738-e747. doi: 10.1097/j.pain.0000000000002470. Epub 2021 Sep 2. PMID 34490850